CLINICAL TRIAL: NCT02662153
Title: Incidence and Predictors of Opioid Overdose and Death Among Users of Opioid Analgesics as Measured by Diagnoses and Death Records - a Retrospective Database Study
Brief Title: Incidence and Predictors of Opioid Overdose and Death Among Long-Term Users of Opioid Analgesics
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: Kaiser Permanente (Other); HealthCore, Inc. (Industry); Vanderbilt University (Other); World Health Information Science Consultants, LLC (Other); Optum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-2; Study 3033-2 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long-term opioid-use cohort: Persons who have received 70 or more days of Schedule II opioid dispensed in a 90-day period, after at least 183 days with no opioid dispensing.
  Interventions: Other: Observation only
- IR/SA to ER/LA Switchers: Persons who have switched to or added on an ER/LA product after stable use of an IR/SA opioid regimen.
  Interventions: Other: Observation only
- IR/SA to IR/SA Switchers: Persons who have switched to or added on a new IR/SA opioid after stable use of a different IR/SA opioid regimen.
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — No intervention.

SUMMARY:
Retrospective study to assess incidence and predictors of opioid abuse overdose and death associated with opioid overdose among patients prescribed opioid products in long-term use.

DETAILED DESCRIPTION:
The purpose of this study is to quantify risk, and predictors of risks for opioid overdose and for death associated with opioid overdose in persons who are or have been long-term recipients of prescriptions for Schedule II opioids. The study uses coded terms in large heath databases maintained by healthcare providers and health insurers, supplemented by overdose deaths identified from the National Death Index. The terms for overdose are combined following validated rules as developed in companion studies. The study is being conducted in parallel with a prospective questionnaire-based cohort study of the same risks.

ELIGIBILITY:
Inclusion Criteria:

* In the primary analysis, persons known to have had at least six months of no opioid dispensing who subsequently receive at least 70 days of Schedule II opioid dispensed within a 90-day period and who have not previously experienced an opioid overdose.
* In a secondary analysis, persons who have been long-term users of IR/SA opioids and who switch to a different Schedule II IR/SA opioid product or to an ER/LA opioid
* In another secondary analysis, persons with at least six months of presence in the health insurance data who have not received opioids in the preceding 30 days, and have not previously experienced an opioid overdose

Exclusion Criteria:

• Experience of opioid overdose in the six months preceding inclusion

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source populations will be those members of the selected health plans and insurance programs identified for which full demographic, provider, facility and pharmacy data are available, and in which protected health information (PHI) can be linked to death certificate information.
  The four large healthcare systems that have established electronic databases for studying coded terminology outcomes selected for this study are: Kaiser Permanente Northwest; HealthCore, Inc. with access to commercial insurance data; Optum with access to commercial insurance data; and Vanderbilt University with access to Medicaid data for the State of Tennessee.
Sampling Method: Non-Probability Sample
Enrollment: 808455 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Opioid overdose - fatal and nonfatal | Retrospective review over period from October 1, 2006 to December 31, 2017
  Opioid overdose as identified in insurance claims, electronic medical records and National Death Index records.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Petronis, Study Chair — Epi Ideas LLC; John D Seeger, Principal Investigator — Optum, Inc.
Locations (4):
- United States (4):
  - HealthCore Inc, Wilmington, Delaware
  - Optum, Boston, Massachusetts
  - Kaiser Permanente Northwest, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee